CLINICAL TRIAL: NCT03281135
Title: Optimizing Cervical Cancer Screening Modalities and Identifying the Molecular Epidemiology of Human Papilloma Virus in Ethiopia: A Cluster Randomized Trial
Brief Title: Optimizing Cervical Cancer Screening Modalities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Addis Ababa University (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Muluken Gizaw Turago, Assistant Professor, Addis Ababa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 058/17/SPH
Record Dates: First submitted 2017-09-08; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer screening; Adherance; HPV typing; HDSS; Ethiopia
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: A cluster randomized trial will be conducted in the Health and Demographic Surveillance Site (HDSS) of Addis Ababa University, School of Public Health which is located in Butajira district. The study population consists of women aged 30-49 who are found among the catchment population of ten Kebele's(Smallest Administrative Unit). Each Kebele will have 2 or more clusters based on the community health workers structure and size. A total of 22 clusters will then be randomized in to two arms. A total of 1760 women will be grouped in to 22 clusters, each comprises 80 women.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV testing (Other): This is an experimental arm for the primary outcome, 'adherence to the procedures'. In this group self sampling will be done using the Evalyn brush for HPV testing.
  Interventions: Other: HPV testing
- Standard care: VIA screening (No Intervention): Control Arm, in which women's are invited to cervical cancer screening as per standard Ethiopian cervical cancer prevention and control guideline. Uptake of screening in this group will be compared with the HPV testing arm group to test for significant differences in adherence.

INTERVENTIONS:
Other: HPV testing — Clusters randomly allocated to this arm of the study will be sensitized to be showed up in nearby health posts for self sampling with Evalyn brush for HPV testing.
  Arms: HPV testing

SUMMARY:
This project aims to optimize cervical cancer screening adherence comparing Arm A (VIA) and Arm B self-sampled Human Papilloma Virus (HPV) testing and determine the molecular epidemiology of HPV, persistence level and identify factors responsible for persistence, and also characterizing the potential dysplasia by biomarkers that describe the disease stage in a population of Ethiopia.

A cluster-randomized trial will be used in this study. The total number of ten kebele's(Smallest administrative unit) will be randomly classified in to two arms(VIA and HPV+VIA).Community health workers will be used as a cluster for randomization. Community sensitization and awareness creation will be performed at health facilities and in communities at social, business or religious gatherings, about cervical cancer and its prevention for eligible women in both arms. Women will be educated about cervical cancer and advice for testing at the Hospital offering VIA (arm A). Women will also be instructed to undergo HPV self-sampling at nearby health posts with a vaginal evalyn brush (arm B). All eligible women on each cluster will be included in the study at both arms. Based on the community health workers number and structure study area there will be about 22 clusters with 80 eligible women on each cluster. Brushes will be sent to the Microbiology Laboratory of Department of Microbiology,Immunology and Parasitology,College of Health Sciences, Addis Ababa University, Addis Ababa, where the laboratory service is sated-up . Trained Microbiologists will perform the laboratory analysis at the HPV laboratory. Only women with samples positive for high-risk HPV (hrHPV) will be contacted and informed to go to the Hospital offering VIA. Further tests will also be performed from the brushes at the collaborators' HPV laboratory, Germany to better characterize the dysplesia.

The women found positive for VIA or hrHPV+VIA will receive cryo treatment at Butajira Hospital. To evaluate the long-term effect and factors for persistence, all eligible women within the catchment area will be visited after 2 years door to-door and asked for a vaginal self-sample and HPV-genotype test. The impact of intervention, factors associated with HPV infection, persistence, clearance, and adherence to the screening service will be seen.

DETAILED DESCRIPTION:
Cervical cancer is the second most common cancer in women worldwide but the commonest in developing countries. In Ethiopia, cervical cancer is the leading cause of morbidity and mortality from all cancers. The Human Papilloma Viruses (HPV) is a necessary cause for cervical cancer (CC). HPVs 16, 18, 31, 33, 35 and 39 are considered as high risk types which are mainly responsible in cervical carcinogenesis.

In developing countries, including Ethiopia, almost all women with cancers present to health care facilities at late stages with advanced disease and poor prognosis. Unlike other reproductive health cancers, cervical cancer can be prevented and even possible to be cured if identified in its early stages. Currently cervical cancer screening by visual inspection with acetic acid (VIA) and immediate treatment with cryotherapy is recommended by World Health Organization(WHO) for low and middle income countries as this method does not require especially trained professionals and more resources and results are available immediately which reduces the attrition rate. However, yet accessing VIA is difficult for many rural women as the service is only available at least at district Hospital level in very few places. Although VIA is accepted by the government in many low income countries, training , maintaining quality assurance, the invasiveness of a pelvic examination and user variability of the test remain critical barriers. Moreover, the short comings of this method includes having of low positive predictive value and lack of evidence on periodic screening performance.

Detection of High risk Human Papilloma Viruses (HrHPV) in the cervix has been recommended in settings wherever possible. World Health Organization (WHO) primarily recommends the HPV test which is very sensitive and a convenient molecular test for cervical cancer screening. This approach is found to be less examiner-dependent, reduce the burden in health system, enhance the accuracy, efficiency and reduce cultural barriers. Therefore, HPV test might be a future option in low and middle income countries.

In Ethiopia, screening with VIA followed by cryotherapy started in 2009 first for women with HIV in selected 14 hospitals and subsequently the service was expanded to 10 additional health institution. Currently the federal ministry of health in Ethiopia has scaled up the service to the general public into public health facilities. However, still majority of women in Ethiopia are residing in rural area where access to screening and treatment facilities is limited or lacking.

So far few studies have been conducted in African settings for assessing the uptake and acceptability of independent screening approaches. Study in Sub Saharan Africa reported higher acceptance of HPV based cervical cancer screening than visual inspection with acetic acid. In Ethiopia there is no adequate information on women uptake, acceptability, adherence and potential barriers of cervical cancer screening for different screening modalities. Moreover, data on HPV prevalence and genotype distribution are rare.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 30 and 49

Exclusion Criteria:

* women with History of hysterectomy or cervical cancer, pregnant women, not meet the eligibility criteria and unable to give consent.

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1760 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Adherence to the procedures | With in 1 year period
  Proportions of women who adhered in the screening and subsequent follow up based on HPV testing using self-sampling versus an offer of attending for a VIA.
  This will be compared based on: A women who accessed the HPV self sampling at health post and accessed VIA and treated for positive result plus untreated for negative result divided by the eligible women in the arm versus A women who accessed the VIA at health facility and treated for positive result plus untreated for negative result divided by the eligible women in the arm.

SECONDARY OUTCOMES:
Number of women that participate in Cervical Cancer Screening in the control (VIA) compared with the number of women that participate in the intervention(Self sampling HPV testing) | With in 1 year period
  This will be measured based on the number of women who attended only the screening procedure after the first sensitization program
Demographic and socio cultural factors associated with uptake and adherence of two different cervical cancer screening procedures | With in 1 year period
  Here we will try to identify and explore socio economic and cultural barriers related with each screening approach.
HPV genotypes among rural women | With in 1 year period
  We will identify HPV genotypes from all collected samples of the study population. Samples will be collected from the community and analyzed centrally in Addis Ababa.

IPD SHARING:
Plan to Share IPD: Undecided
We will see

REFERENCES:
- [Derived] Teka B, Gizaw M, Firdawoke E, Addissie A, Sisay TA, Schreckenberger C, Skof AS, Thies S, Mihret A, Kantelhardt EJ, Abebe T, Kaufmann AM. A Technical Comparison of Human Papillomavirus Genotyping Assays from a Population-Based Cervical Cancer Screening in South Central Ethiopia. Cancer Manag Res. 2022 Jul 29;14:2253-2263. doi: 10.2147/CMAR.S360712. eCollection 2022. PMID 35937937